CLINICAL TRIAL: NCT01888367
Title: A Randomized, Blinded, Placebo and Standard of Care Controlled Efficacy, Safety, and Tolerability Study of up to 20 mL of DFA-02 in Patients Undergoing Abdominal Surgery
Brief Title: Safety, Efficacy and Tolerability Study of up to 20 mL of DFA-02 in Patients Undergoing Abdominal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DFA-02-CD-005
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Surgical Site Infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DFA-02 Antibiotic Gel (Experimental): Up to 20 mL of DFA-02 antibiotic gel will be placed in the surgical incision after closure of the fascia and before skin closure.
  Interventions: Drug: DFA-02 Antibiotic Gel
- DFA-02 Placebo Gel (Placebo Comparator): Up to 20 mL of DFA-02 placebo gel will be placed in the surgical incision after closure of the fascia and before skin closure.
  Interventions: Drug: DFA-02 Placebo Gel
- Standard of Care (No Intervention): Prior to final closure of the surgical incision, the incision will be irrigated with normal saline and no gel will be applied.

INTERVENTIONS:
Drug: DFA-02 Antibiotic Gel
  Arms: DFA-02 Antibiotic Gel
Drug: DFA-02 Placebo Gel
  Arms: DFA-02 Placebo Gel

SUMMARY:
This is a randomized, blinded, placebo and standard of care controlled study of the efficacy of a novel antibiotic containing gel compared to placebo gel in preventing surgical site infection after abdominal surgery. patients will be randomized to active or placebo gel in a double-blind manner. The gel will be applied a single time in the incision during closure at the end of surgery. A cohort of patients will also be randomized to standard of care, saline irrigation at prior to skin closure, in an open manner. The efficacy, safety and tolerability of the active gel will be assessed compared to the control group (combined placebo gel and standard of care groups). Patients will be randomized to DFA-02 active gel: placebo gel: standard of care in a 4:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older;
2. If female, the subject must be postmenopausal, surgically sterilized or, if of child-bearing potential, she must have a negative serum or urine pregnancy test within 48 hours of surgery and agree to use adequate birth control during the study and for 30 days after the administration of study agent;
3. Body mass index (BMI) ≥ 20;
4. Scheduled to undergo non-emergent abdominal surgery involving a planned incision of 7 cm or greater;
5. Willing and able to give informed consent;
6. Available for evaluation from Baseline until final evaluation at 30 days post-surgery.

Exclusion Criteria:

1. Known hypersensitivity to gentamicin, vancomycin, other aminoglycoside antibiotics or the excipients of the study products;
2. Emergency surgery;
3. Significant concomitant surgical procedure;
4. Prior laparotomy within the last 60 days of the planned procedure;
5. Planned second laparotomy or abdominal surgical procedure within 30 days of the planned first procedure;
6. Expectation that a surgical drain will be placed in the incision;
7. Preoperative sepsis, severe sepsis, or septic shock;
8. Abdominal wall infection/surgical site infection from previous laparotomy/laparoscopy or for any reason;
9. Active systemic infection or systemic (oral or intravenous) antibiotic therapy within the 1 week prior to the date of surgery other than specified preoperative antimicrobial prophylaxis;
10. Requirement for gentamicin or vancomycin preoperative antimicrobial prophylaxis;
11. Concurrent systemic use of other potentially neurotoxic, nephrotoxic, and/or ototoxic drugs;
12. Preoperative evaluation suggesting an intra-abdominal process that might preclude full closure of the skin;
13. Ongoing treatment (e.g. chemotherapy, radiation) for non-colorectal cancer;
14. History of significant drug or alcohol abuse;
15. Serum Creatinine > 1.8 mg/dL;
16. Serum Bilirubin > 2.5 times upper limit of normal;
17. Subjects who are immunocompromised including but not limited to systemic corticosteroid use or chemotherapy/radiation during the 30 days prior to surgery, organ transplantation, or HIV infection;
18. Known history of HIV;
19. Pregnant or lactating, or if of childbearing potential not practicing a birth control method with a high degree of reliability;
20. Refusal to accept medically indicated blood products;
21. Participation within 30 days before the start of this study in any experimental drug or device study, or currently participating in a study in which the administration of investigational drug or device within 60 days is anticipated;
22. Unable to participate in the study for any reason in the opinion of the Principal Investigator;
23. Postsurgical life expectancy of less than 30 days;
24. Expected discharge from the hospital less than 3 days after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Bennett-Guerrero, MD, Study Director — Duke Clinical Research Institute
Locations (31):
- United States (31):
  - Florence, Alabama
  - Sheffield, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Laguna Hills, California
  - Los Angeles, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Weston, Florida
  - Columbus, Georgia
  - Powder Springs, Georgia
  - Indianaoplis, Indiana
  - Alexandria, Louisiana
  - New Orleans, Louisiana
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Las Vegas, Nevada
  - Albany, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Bellaire, Texas
  - Nassau Bay, Texas
  - Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Groups:
- DFA-02 Antibiotic Gel: Up to 20 mL of DFA-02 antibiotic gel will be placed in the surgical incision after closure of the fascia and before skin closure.
  DFA-02 Antibiotic Gel
- DFA-02 Placebo Gel: Up to 20 mL of DFA-02 placebo gel will be placed in the surgical incision after closure of the fascia and before skin closure.
  DFA-02 Placebo Gel
Period: Overall Study
Arm/Group | DFA-02 Antibiotic Gel | DFA-02 Placebo Gel | Standard of Care
Started | 296 | 71 | 78
Completed | 288 | 66 | 73
Not Completed | 8 | 5 | 5
Not completed — Physician Decision | 3 | 4 | 2
Not completed — Death | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — 30-Day Visit Too Early (< 28 Days) | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFA-02 Antibiotic Gel | DFA-02 Placebo Gel | Standard of Care | Total
Number analyzed (Participants) | 296 | 71 | 78 | 445
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (14.6) | 58.8 (15.7) | 59.6 (14.7) | 59.8 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 33 | 45 | 220
  Male | 154 | 38 | 33 | 225
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 8 | 1 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 31 | 10 | 4 | 45
  White | 255 | 60 | 74 | 389
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 296 | 71 | 78 | 445

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Surgical Site Infections
Time Frame: Within 30 days of surgery
Population: The number of SSIs from the day of surgery to 30 days post-op could only be assessed in the 427 completed patients. Central adjudication by the Clinical Events Committee was not able to assess the presence or absence of SSI for two patients, one in the DFA-02 group and one in the SOC group so the total analyzed is only 425.
Measure: Number; unit: participants
Arm/Group | DFA-02 Antibiotic Gel | DFA-02 Placebo Gel | Standard of Care
Number analyzed (Participants) | 287 | 66 | 72
participants | 42 | 14 | 25

2. Secondary Outcome: Number of Patients With Adverse Events
Time Frame: Within 30 days of surgery
Population: The safety analysis was "as treated". For 4 patients the actual treatment given could not be assigned due to conflicting data excluding them from the analysis leaving 441 subjects out of the 445 randomized. The DFA-02 Gel and Placebo Gel groups were decreased as the patients who did not receive gel were counted in the SOC group.
Measure: Number; unit: participants
Arm/Group | DFA-02 Antibiotic Gel | DFA-02 Placebo Gel | Standard of Care
Number analyzed (Participants) | 284 | 64 | 93
participants | 267 | 61 | 86

3. Secondary Outcome: Change in Serum Creatinine Measurements From Baseline
Description: Change from baseline in micromoles/liter
Time Frame: Within 4 days of surgery
Population: 402 of the 445 patients had both baseline and post-operative creatinine measurements. Safety analyses were "as treated" so patients randomized to gel but did not receive it in surgery were counted in the SOC group.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | DFA-02 Antibiotic Gel | DFA-02 Placebo Gel | Standard of Care
Number analyzed (Participants) | 262 | 61 | 79
micromoles/liter | -10.2 (18.2) | -9.9 (12.8) | -10.2 (27.0)

4. Secondary Outcome: Cumulative ASEPSIS Score for Each Patient
Description: Total ASEPSIS score with a range of 0-65 points with lower scores being better. The score is the sum of: Antibiotic Use (10 points), Drainage of Pus Under Local Anesthesia (5 points), Debridement Under General Anesthesia (10 points), Serous Discharge (5 points), Erythema (5 points), Purulent Exudate (5 points), Separation of Deep Tissues (10 points) and Isolation of Bacteria from Discharge (10 points). Source: Wilson AP, Treasure T, Sturridge MF, Gruneberg RN. Lancet. 1986:1(8476):311-3.
Time Frame: Through post-operative Day 4
Population: Safety analyses were "as treated" so patients who were randomized to gel but did not receive it are counted as SOC. For 4 patients, the actual treatment given could not be assigned due to conflicting data excluding them from the analysis leaving 441 subjects out of the 445 randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DFA-02 Antibiotic Gel | DFA-02 Placebo Gel | Standard of Care
Number analyzed (Participants) | 284 | 64 | 93
units on a scale | 17.5 (8.1) | 18.5 (3.5) | 23.0 (3.5)

ADVERSE EVENTS:
Time Frame: From time of surgery until 30 days post-op.
Description: Subjects queried at each visit for any potential adverse events. The safety analysis was "as treated". For 4 patients the actual treatment given could not be assigned due to conflicting data excluding them from the analysis leaving 441 subjects out of the 445 randomized. The DFA-02 Gel and Placebo Gel groups were decreased as the surgeon did not administer the gel to all patients randomized to gel. Those patients were counted in the SOC group.
Arm/Group | DFA-02 Antibiotic Gel | DFA-02 Placebo Gel | Standard of Care
Serious Adverse Events (participants affected / at risk) | 59/284 | 14/64 | 21/93
Other Adverse Events (participants affected / at risk) | 267/284 | 61/64 | 86/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFA-02 Antibiotic Gel (N=284) | DFA-02 Placebo Gel (N=64) | Standard of Care (N=93)
Pelvic Abscess (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Pneuomia (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abdominal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hematoma Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Incision Site Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Splenic Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subdiaphragmatic Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Small Intestine Obstruction (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Enterocutaneous Fistula (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Abdominal Wall Hematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Localized Abdominal Fluid Collection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 7 (7) | 2 (2) | 4 (4)
Anastomotic Leak (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anastomotic Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bladder Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative Renal Failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound Secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 1 (1)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device Dislocation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFA-02 Antibiotic Gel (N=284) | DFA-02 Placebo Gel (N=64) | Standard of Care (N=93)
Procedural Pain (Injury, poisoning and procedural complications) | 143 (143) | 32 (32) | 52 (52)
Procedural Nausea (Injury, poisoning and procedural complications) | 28 (28) | 8 (8) | 10 (10)
Anemia Postoperative (Injury, poisoning and procedural complications) | 26 (26) | 6 (6) | 12 (12)
Incision Site Pain (Injury, poisoning and procedural complications) | 17 (17) | 3 (3) | 3 (3)
Postoperative Ileus (Injury, poisoning and procedural complications) | 12 (12) | 3 (3) | 4 (4)
Seroma (Injury, poisoning and procedural complications) | 12 (12) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 118 (118) | 32 (32) | 41 (41)
Vomiting (Gastrointestinal disorders) | 39 (39) | 15 (15) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 25 (25) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 17 (17) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 14 (14) | 4 (4) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 10 (10) | 3 (3) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 46 (46) | 8 (8) | 18 (18)
Hypokalemia (Metabolism and nutrition disorders) | 43 (43) | 7 (7) | 17 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 39 (39) | 9 (9) | 14 (14)
Hypocalcemia (Metabolism and nutrition disorders) | 37 (37) | 7 (7) | 15 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 25 (25) | 5 (5) | 12 (12)
Hypoproteinemia (Metabolism and nutrition disorders) | 26 (26) | 4 (4) | 10 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 28 (28) | 2 (2) | 8 (8)
Hyponatremia (Metabolism and nutrition disorders) | 19 (19) | 4 (4) | 8 (8)
Hypochloremia (Metabolism and nutrition disorders) | 14 (14) | 1 (1) | 5 (5)
Urine Output Decreased (Investigations) | 26 (26) | 5 (5) | 10 (10)
Oxygen Saturation Decreased (Investigations) | 16 (16) | 3 (3) | 6 (6)
Amylase Decreased (Investigations) | 3 (3) | 0 (0) | 5 (5)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 28 (28) | 7 (7) | 3 (3)
Incision Site Infection (Infections and infestations) | 17 (17) | 3 (3) | 4 (4)
Pelvic Abscess (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 30 (30) | 6 (6) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 42 (42) | 9 (9) | 15 (15)
Tachycardia (Cardiac disorders) | 46 (46) | 14 (14) | 15 (15)
Leukocytosis (Blood and lymphatic system disorders) | 29 (29) | 6 (6) | 12 (12)
Anemia (Blood and lymphatic system disorders) | 24 (24) | 4 (4) | 10 (10)
Hematuria (Renal and urinary disorders) | 12 (12) | 8 (8) | 8 (8)
Urinary Retention (Renal and urinary disorders) | 14 (14) | 4 (4) | 9 (9)
Hypertension (Vascular disorders) | 34 (34) | 7 (7) | 6 (6)
Hypotension (Vascular disorders) | 23 (23) | 2 (2) | 9 (9)
Anxiety (Psychiatric disorders) | 19 (19) | 2 (2) | 7 (7)
Insomnia (Psychiatric disorders) | 15 (15) | 2 (2) | 9 (9)
Headache (Nervous system disorders) | 17 (17) | 3 (3) | 5 (5)

LIMITATIONS AND CAVEATS:
The number of culture positive SSIs were too small to draw any conclusions on antibiotic resistance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less